CLINICAL TRIAL: NCT04349241
Title: Efficacy and Safety of Favipiravir in Management of COVID-19
Acronym: FAV-001
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hany Dabbous, Assistant professor of Faculty of Medicine, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU P14 / 2020
Record Dates: First submitted 2020-04-13; First posted 2020-04-16 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Coronavirus Disease (COVID-19)
MeSH Terms: conditions — COVID-19 | interventions — favipiravir

STUDY DESIGN:
Intervention Model Description: A block-randomization scheme will be generated by computer software. 100 patients with confirmed COVID-19 will be randomized between favipiravir and the standard of care therapy (treated according to the national protocol) in a 1:1 ratio.
  Group 1: 50 patients will receive the investigational drug favipiravir. Group 2: 50 patients will receive oseltamivir and hydroxychloroquine as the national standard of care therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- favipiravir (Experimental): favipiravir in a regimen of 3200 mg (1600 mg 12 hourly) loading dose on day-1 followed by 1200 mg maintenance dose (600 mg 12 hourly daily) on day-2 to day-10
  Interventions: Drug: favipiravir
- Standard of care therapy (Active Comparator): oseltamivir 75 mg 12 hourly for 5-10 days and hydroxychloroquine 400mg 12 hourly day -1 followed by 200mg 12 hourly daily on day- 2 to day-5-10.
  Interventions: Drug: Standard of care therapy

INTERVENTIONS:
Drug: favipiravir — pyrazine carboxamide derivative (6-fluoro-3-hydroxy-2-pyrazinecarboxamide), a new type of RNA-dependent RNA polymerase (RdRp) inhibitor
  Other Names: pyrazine carboxamide derivative
  Arms: favipiravir
Drug: Standard of care therapy — oseltamivir 75 mg 12 hourly for 5-10 days and hydroxychloroquine 400mg 12 hourly day -1 followed by 200mg 12 hourly daily on day- 2 to day-5-10
  Other Names: National Egyptian guideline
  Arms: Standard of care therapy

SUMMARY:
Randomized controlled interventional trial (Clinical Trial) phase 3 to assess the safety and efficacy of favipiravir versus the standard care therapy in the treatment of patients with COVID-19.

DETAILED DESCRIPTION:
Study Procedures:

Screening phase:

* Obtaining an informed consent

  * Written signed and dated informed consent will be obtained from each patient before being entered into the study. The investigator, or a person designated by the investigator, should fully inform the subject or, if the subject is unable to provide informed consent, the subject's legally acceptable representative, of all pertinent aspects of the trial. This will be obtained from each subject in accordance with the recommendation of the revised Declaration of Helsinki. The investigator will explain the nature, purpose and risks of the study. It will be clearly stated that the patient is free to withdraw from the study at any time for any reason without prejudice to future care, and with no obligation to give the reason for withdrawal.
  * In case the patient is unable to provide his/her consent the legal guardian will give verbal approval on behaves of the patient and after he he/she will be well informed by the study design, procedure, risk and benefits over phone call.
  * If it is difficult to reach the legal guardian, emergency approval will be obtained by Professional Legal Representative who will be the head authorities of the isolation hospital.
* Full medical history, concurrent medications, demographic data will be obtained.
* A thorough physical examination will be performed.
* Body weight, height, BMI, vital signs (blood pressure, heart rate and temperature) and Blood oxygen saturation) will be recorded.
* Chest X-ray or CT chest will be recorded.
* Laboratory to perform the following tests:

Complete blood count with differential counts, COVID -19 PCR test by nasopharyngeal swab. C-reactive protein and serum ferritin level. Renal function tests (RFTs) (serum creatinine), Liver function tests (LFTs) (alanine amino transferase (ALT), aspartate amino transferase (AST), total and direct bilirubin), Coagulation test; prothrombin time and INR. HIV antibody, HCV antibody and HBV surface antigen (HBsAg). Urine pregnancy test for females.

Treatment phase for eligible patients:

* Eligibility confirmed
* The patient will receive information regarding the treatment duration, how to take the study treatment and the dose of the study treatment.
* The patient will receive information regarding the identification and notification of adverse events as diarrhea that occurs in about 25 % of patients and mild elevation of transaminases.
* The patient will be advised to record the daily dosing of study medications that were taken in diaries. If the patient is fatigued or uneducated the clinical pharmacist or the treating physician will be responsible for recording.
* Concomitant medications will also be recorded.
* Eligible patients in group 1 will be given favipiravir in a regimen of 3200 mg (1600 mg 12 hourly) loading dose on day-1 followed by 1200 mg maintenance dose (600 mg 12 hourly daily) on day-2 to day-10.
* Eligible patients in group 2 will receive oseltamivir 75 mg 12 hourly for 5-10 days and hydroxychloroquine 400mg 12 hourly day -1 followed by 200mg 12 hourly daily on day- 2 to day-5-10.
* Clinical assessment will be performed on days 3 and 7 and adverse events will be recorded.
* Laboratory follow up: Days 3 and 7 of treatment

  * Liver function tests (ALT and AST).
  * COVID -19 PCR test by nasopharyngeal swab.
  * C-reactive protein and serum ferritin levels. End point of the study: Day 14 assessment
* The patient's health status and the presence of adverse events will be assessed.
* Complete physical examination.
* Vital signs (blood pressure, heart rate and temperature) will be recorded.
* Follow-up CXR and /or CT scan.
* Liver function tests (LFTs) (alanine amino transferase (ALT), aspartate amino transferase (AST), total and direct bilirubin).
* C-reactive protein and serum ferritin level.
* COVID -19 PCR test by nasopharyngeal swab
* Post treatment period up to 30 days after end of treatment:
* Vital signs (blood pressure, heart rate and temperature) will be recorded.
* Symptoms and signs assessment will be done.

ELIGIBILITY:
Inclusion Criteria:

Patients aged between 18 and 80 years.

Patients with confirmed COVID-19 documented by a diagnostic laboratory test (e.g., nasopharyngeal swab) at the time of illness.

And Have mild to moderate symptoms according to the national protocol classification of patients.

Exclusion Criteria:

Patients have severe or immediately life-threatening COVID-19, Severe disease is defined as: dyspnea, respiratory frequency ≥ 30/min, blood oxygen saturation ≤ 93%, partial pressure of arterial oxygen to fraction of inspired oxygen ratio < 300, and/or lung infiltrates > 50% within 24 to 48 hours Life-threatening disease is defined as: respiratory failure, septic shock, and/or multiple organ dysfunction or failure

Pregnant or lactating females.

Participation in any investigational clinical study, other than observational, within the past 30 days; or plans to participate in such a study at any time from the day of enrollment until 30 days post-treatment in the current study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-04-18 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-20 (Actual)

PRIMARY OUTCOMES:
Viral clearance | 14 days
  Two successive negative COVID-19 PCR analysis tests 48-72 hours apart
Clinical improvement | 14 days
  Normal body temperature for 48 hours

SECONDARY OUTCOMES:
Radiological Improvement | 14 days
  Improvement of radiological abnormalities at day 14

CONTACTS AND LOCATIONS:
Overall Officials: Hany Dabbous, Principal Investigator — Ain Shams University
Locations (1):
- Faculty of Medicine Ain Shams University Research Institute- Clinical Research Center, Cairo, Non-US, Egypt

IPD SHARING:
Plan to Share IPD: No